CLINICAL TRIAL: NCT05696418
Title: Effect of Using Mobile Bearing on the Incidence Rate of Anterior Knee Pain in Primary Total Knee Arthroplasty Without Patellar Resurfacing (A Randomized Controlled Clinical Trial)
Brief Title: Anterior Knee Pain in Mobile Bearing Versus Fixed Bearing in TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDMS-Orthopedics-2-2023
Record Dates: First submitted 2023-01-11; First posted 2023-01-25 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Joint Diseases; Arthritis Knee; Arthroplasty Complications
Keywords: Mobile bearing; Fixed bearing; Knee Arthroplasty
MeSH Terms: conditions — Joint Diseases | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mobile Bearing Design TKA (Experimental): Patients who were randomized to receive the PFC Sigma Mobile Bearing TKA system
  Interventions: Procedure: Total knee arthroplasty with a Mobile Bearing system.
- Fixed Bearing Design TKA (Experimental): Patients who were randomized to receive the PFC Sigma Fixed Bearing TKA system
  Interventions: Procedure: Total knee arthroplasty with a Fixed Bearing system.

INTERVENTIONS:
Procedure: Total knee arthroplasty with a Mobile Bearing system. — The prostheses will be cruciate scarifying cemented DePuy Synthes PFC Sigma with a Mobile Bearing system without resurfacing the patella.
  Arms: Mobile Bearing Design TKA
Procedure: Total knee arthroplasty with a Fixed Bearing system. — The prostheses will be cruciate scarifying cemented DePuy Synthes PFC Sigma with a Fixed Bearing system without resurfacing the patella.
  Arms: Fixed Bearing Design TKA

SUMMARY:
Osteoarthritis is the most common cause of chronic joint disease, and its incidence has increased due to the high average life expectancy, in addition to the high incidence of obesity. Total knee arthroplasty is currently an accepted treatment for severe degenerative conditions and there are various implant systems with special features depending on component geometry, degree of fit of the articular surfaces, and fixation techniques. A tibial component with mobile polyethylene has been developed as an alternative to fixed polyethylene because it has theoretical advantages in terms of increasing the range of motion, reducing wear conditions, and reducing the incidence of anterior knee pain when the articular surface of the patella is not resurfaced.

DETAILED DESCRIPTION:
The study is a randomized controlled clinical trial where the sample will be collected within one year from the date of approval of the Scientific Research Council at Damascus University. The sample consists of patients undergoing a total primary knee arthroplasty without patellar resurfacing following primary arthritis knee. The patients will be randomly divided into two groups. The first will be a primary total knee arthroplasty with a mobile bearing, and the second group with a fixed bearing. Then the patients will be followed for at least one year.

The data of the patients included in the study will be collected before the surgical operation, then the surgery; followed up for at least one year after it, and then compared between the two groups in terms of a range of motion and functional and clinical results according to the Knee Society Score (KSS) and the anterior knee pain scale, and patient satisfaction assessment according to the Forgotten Joint Scale (FJS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with expected primary total knee arthroplasty

Exclusion Criteria:

* Mediolateral instability
* Infective arthritis
* Severe deformity
* Revision
* Patients with severe obesity according to the Body Mass Index (BMI < 35).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Anterior knee pain | 1-2 years after surgery
  Anterior knee pain will be assessed by questionnaire.

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 1-2 years after surgery
  Clinical and functional outcomes will be assessed by Knee Society Score (KSS). The knee society score (KSS) contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag. The Knee Society Score is divided into three sessions: it consists of the Knee Score (100 points), the Knee Function (100 points), and the patient classification system. The classification system separates the patients into three categories depending on their medical conditions - A: unilateral or bilateral (contralateral knee operated successfully); B: unilateral -contralateral knee symptomatic; C: multiple arthritis. The two scores are initially marked at zero and points are assigned or deducted according to specific criteria.
Forgotten Joint Scale (FJS) | 1-2 years after surgery
  Patient satisfaction will be assessed by Forgotten Joint Scale (FJS). The FJS-12 consists of twelve equally-weighted questions that are each answered on a five-level Likert scale aimed to measure patient satisfaction. The questionnaire was developed with the consideration that joint awareness is a very important and highly discriminative outcome parameter, especially in patients with good-to-excellent joint function. Answers to each question are individually scored and summed to create a raw composite score that is normalized to range from 0 (worst condition) to 100 points (best condition)
perioperative complications | assessed within two weeks intervals until 6 months after surgery
  such as infection, VET, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jaber Ibrahim, M.D, Ph.D, Study Director — Damascus University
Locations (1):
- Damascus university, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang CH, Ma HM, Lee YM, Ho FY. Long-term results of low contact stress mobile-bearing total knee replacements. Clin Orthop Relat Res. 2003 Nov;(416):265-70. doi: 10.1097/01.blo.0000093890.12372.46. PMID 14646769
- [Background] Kim YH, Kook HK, Kim JS. Comparison of fixed-bearing and mobile-bearing total knee arthroplasties. Clin Orthop Relat Res. 2001 Nov;(392):101-15. doi: 10.1097/00003086-200111000-00013. PMID 11716371
- [Background] Dennis DA, Komistek RD, Scuderi GR, Zingde S. Factors affecting flexion after total knee arthroplasty. Clin Orthop Relat Res. 2007 Nov;464:53-60. doi: 10.1097/BLO.0b013e31812f785d. PMID 17621230
- [Background] Hooper G, Rothwell A, Frampton C. The low contact stress mobile-bearing total knee replacement: a prospective study with a minimum follow-up of ten years. J Bone Joint Surg Br. 2009 Jan;91(1):58-63. doi: 10.1302/0301-620X.91B1.20484. PMID 19092005
- [Background] Li B, Bai L, Fu Y, Wang G, He M, Wang J. Comparison of clinical outcomes between patellar resurfacing and nonresurfacing in total knee arthroplasty: retrospective study of 130 cases. J Int Med Res. 2012;40(5):1794-803. doi: 10.1177/030006051204000517. PMID 23206460
- [Background] Khan A, Pradhan N. Results of total knee replacement with/without resurfacing of the patella. Acta Ortop Bras. 2012;20(5):300-2. doi: 10.1590/S1413-78522012000500011. PMID 24453622
- [Background] Waters TS, Bentley G. Patellar resurfacing in total knee arthroplasty. A prospective, randomized study. J Bone Joint Surg Am. 2003 Feb;85(2):212-7. doi: 10.2106/00004623-200302000-00005. PMID 12571296
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572